CLINICAL TRIAL: NCT00871104
Title: Evaluation of the Efficacy and Safety of Fosfomycin Plus Imipenem for the Treatment of Methicillin-resistant Staphylococcus Aureus (MRSA) Infective Endocarditis.
Brief Title: Fosfomycin Plus Imipenem for Treatment of Infective Endocarditis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOSIMI; EudraCT number: 2008-008683-28
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Fosfomycin; Imipenem; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): IV fosfomycin and imipenem adjusted to renal function
  Interventions: Drug: Fosfomycin and imipenem
- 2 (Active Comparator): IV Vancomycin twice a day with valley leves higher than 15 mcg/kg
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fosfomycin and imipenem — IV Fosfomycin 2 gr./6 hours and IV Imipenem 1 gr./6 hours adjusted acoording to renal function during 4-8 weeks
  Arms: 1
Drug: Vancomycin — IV Vancomycin 30 mg/kg twice a day with valley leves higher than 15 mcg/kg
  Arms: 2

SUMMARY:
The study evaluates the efficacy and safety of fosfomycin and imipenem for the treatment of methicillin-resistant staphyloccocus aureus infective endocarditis in comparison to vancomycin, the standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Suspected methicillin-resistant staphyloccocus aureus infective endocarditis on a native valve, prosthetic valve or pacemakers´s electrode or defibrillators with definitive or probable diagnosis by the modified Duke criteria (Li J, et al. Clin Infect Dis. 2000).
* Patients over 18 years.

Exclusion Criteria:

* Patients who did not sign informed consent.
* Patients with active consumption intravenous drug.
* Patients with emergent surgery criteria (<72 hours).
* Patients or cardiogenic shock.
* Patients with antibiotic active against MRSA over 72 hours or they may need another antibiotic active against MRSA than those in the study.
* Patients with chronic renal failure on hemodialysis who received empirical treatment with vancomycin as a single dose and have a valley ≥ 15 mcg / mL on the third day.
* Patients with MRSA strains resistant to fosfomycin (MIC> 64 mg / L) (<10%) or vancomycin (MIC> 2 mg / L) or with an MIC to vancomycin of 2 mg / L.
* Patients with any formal contraindication to be treated with study drugs
* Patients treated with any investigational drug within 30 days prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2015-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with negative blood cultures. | 7 days

SECONDARY OUTCOMES:
Toxicity due to treatment | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Asunción Moreno Camacho, MD, Principal Investigator — Hospital Clínic of Barcelona
Locations (10):
- Spain (10):
  - Hospital Sant Pau of Barcelona, Barcelona, Catalonia
  - Hospital Clínic of Barcelona, Barcelona, Catalonia
  - Hospital Bellvitge of Barcelona, Barcelona, Catalonia
  - Fundación Hospital Alcorcón, Alcorcón - Madrid, Madrid
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital Virgen Macarena, Seville
  - Hospital Virgen del Rocío, Seville

REFERENCES:
- [Derived] Pericas JM, Hernandez-Meneses M, Munoz P, Martinez-Selles M, Alvarez-Uria A, de Alarcon A, Gutierrez-Carretero E, Goenaga MA, Zarauza MJ, Falces C, Rodriguez-Esteban MA, Hidalgo-Tenorio C, Hernandez-Cabrera M, Miro JM; Spanish Collaboration on Endocarditis-Grupo de Apoyo al Manejo de la Endocarditis Infecciosa en Espana (GAMES). Characteristics and Outcome of Acute Heart Failure in Infective Endocarditis: Focus on Cardiogenic Shock. Clin Infect Dis. 2021 Sep 7;73(5):765-774. doi: 10.1093/cid/ciab098. PMID 33560404
- [Derived] Pericas JM, Ambrosioni J, Munoz P, de Alarcon A, Kestler M, Mari-Hualde A, Moreno A, Goenaga MA, Farinas MC, Rodriguez-Alvarez R, Ojeda-Burgos G, Galvez-Acebal J, Hidalgo-Tenorio C, Noureddine M, Miro JM; GAMES Investigators. Prevalence of Colorectal Neoplasms Among Patients With Enterococcus faecalis Endocarditis in the GAMES Cohort (2008-2017). Mayo Clin Proc. 2021 Jan;96(1):132-146. doi: 10.1016/j.mayocp.2020.06.056. PMID 33413809
- [Derived] Pericas JM, Llopis J, Munoz P, Galvez-Acebal J, Kestler M, Valerio M, Hernandez-Meneses M, Goenaga MA, Cobo-Belaustegui M, Montejo M, Ojeda-Burgos G, Sousa-Regueiro MD, de Alarcon A, Ramos-Martinez A, Miro JM; GAMES Investigators. A Contemporary Picture of Enterococcal Endocarditis. J Am Coll Cardiol. 2020 Feb 11;75(5):482-494. doi: 10.1016/j.jacc.2019.11.047. PMID 32029130
- [Derived] del Rio A, Gasch O, Moreno A, Pena C, Cuquet J, Soy D, Mestres CA, Suarez C, Pare JC, Tubau F, Garcia de la Maria C, Marco F, Carratala J, Gatell JM, Gudiol F, Miro JM; FOSIMI Investigators. Efficacy and safety of fosfomycin plus imipenem as rescue therapy for complicated bacteremia and endocarditis due to methicillin-resistant Staphylococcus aureus: a multicenter clinical trial. Clin Infect Dis. 2014 Oct 15;59(8):1105-12. doi: 10.1093/cid/ciu580. Epub 2014 Jul 21. PMID 25048851